CLINICAL TRIAL: NCT04090333
Title: Endocrinological Profile in Patients With Medication-overuse Headache Before
Brief Title: Endocrinological Profile in Patients With Medication-overuse Headache Before and After Withdrawal Therapy
Acronym: ENDOMOH
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Louise Carlsen, MD, PhD-student, Danish Headache Center
Other Study IDs: H-19023379
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Endocrine Disorder; Deficiency; Medication Overuse Headache; Migraine
MeSH Terms: conditions — Endocrine System Diseases; Headache Disorders, Secondary; Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and urine collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard withdrawal therapy — All painkillers are abruptly stopped for a 2 months period.

SUMMARY:
The project will be conducted to investigate the hormonal homeostasis in men and women, with a special emphasis on sex hormones in men and AMH level in women, before and after withdrawal of the overused analgesics among MOH patients. Additionally, a more broad endocrine profile will be explored before and after withdrawal.

It is hypothesized that patients with MOH have disturbed hormone levels, which is normalized after withdrawal of the medication-overuse.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MOH diagnosis according to the ICHD-III (1).
* Capable of completing headache diary and headache calendar
* Age 18-60 years old for men and 18-50 years old for women
* Signed informed consent
* BMI 19-30

Exclusion Criteria:

* Severe physical illness
* Severe psychiatric disorders requiring pharmacological treatment
* Addiction to alcohol or other drugs
* Pregnancy or breastfeeding
* Menopause, either natural or surgical (only women)
* Inability to provide reliable information about medical history

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients fulfilling the ICHD3-criteria for medication-overuse headache. 50 men and 50 women.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Comparison of levels of following circulating and excreted hormones in the pituitary-gonadal axis at baseline and after 2 months of withdrawal | From baseline to 2 months follow-up
  For male patients with MOH: LH, FSH, testosterone, ratio free testosterone/LH, E2, AMH, inhibin B and sex hormone-binding globulin (SHBG) For female patients with MOH: AMH Standardized reference values are available for all the mentioned levels of sex hormones.

SECONDARY OUTCOMES:
Days with analgesics, migraine medication, rescue medication and other medication during the withdrawal period. | At baseline; and from baseline to 2 months follow-up
Types and doses of analgesics, migraine medication, rescue medication and other medication during the withdrawal period. | At baseline; and from baseline to 2 months follow-up
Levels of circulating pharmaceuticals at baseline and 2 months after withdrawal with special focus on paracetamol, NSAIDs, triptans and opioids for relation to levels of hormones from both genders. | At baseline; and from baseline to 2 months follow-up
Levels of circulating pharmaceutical metabolites (known and potential new unknown) of pa-racetamol, NSAIDs, triptans and opioids at baseline and 2 months after withdrawal with special focus for relation to levels of hormones from both genders. | At baseline; and from baseline to 2 months follow-up
Comparison of a broad screening of the endocrinological profile before and 2 months after withdrawal. | At baseline; and from baseline to 2 months follow-up
Relation between headache days per month and levels of hormones at baseline and at 2 months follow-up. | At baseline; and from baseline to 2 months follow-up
Relation between reproductive health related to compensated hypogonadism, e.g. erectile dysfunction at baseline and at 2 months follow-up. | At baseline; and from baseline to 2 months follow-up
Relation between PSS, HADS, and FSMC, respectively, and levels of sex hormones at baseline and at 2 months follow-up, since hormone levels may be affected in stressed periods | At baseline; and from baseline to 2 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carlsen LN, Nielsen BS, Rouw C, Petersen MR, Lindh CH, Krais AM, Westgate CSJ, Jeppesen JV, Jensen LB, Kristensen SG, Ziebe S, Jensen RH, Kristensen DM. Overuse of analgesics can affect the fertility biomarker Anti-Mullerian Hormone in females. A translational study. Cephalalgia. 2024 Nov;44(11):3331024241290530. doi: 10.1177/03331024241290530. PMID 39558601